CLINICAL TRIAL: NCT05597566
Title: Predictive Effect of Neuroinflammatory Factors on the Efficacy of Modified Electroconvulsive Therapy in the Treatment of Senile Depression Accompanied by Suicidal Ideation
Brief Title: Predictive Effect of Neuroinflammatory Factors of the MECT in Treatment of Senile Depression
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Qinge Zhang (Other)
Responsible Party: Sponsor-Investigator, Qinge Zhang, Professor, Capital Medical University
Organization: Capital Medical University (Other)
Other Study IDs: KM202010025011
Record Dates: First submitted 2022-09-20; First posted 2022-10-28 (Actual); Last update posted 2022-10-28 (Actual); Status verified 2022-10

CONDITIONS: Major Depression Disorder
Keywords: neuroinflammatory factors; modified electroconvulsive therapy(MECT)

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Elderly depression patients with suicidal ideation: Conformity: Age 60-85 years old; meet DSM-5 diagnostic criteria for major depressive disorder; currently in acute phase, HDRS-17 ≥ 24; history of suicide attempt in this depressive episode; current suicidal ideation, SIOSS ≥ 12.Exclusions: Patients with unstable physical diseases; patients currently suffering from acute inflammatory infection or chronic inflammatory disease; participated in another interventional clinical study within the past 1 month; previous or current diagnosis of other psychiatric diseases by DSM-IV ; abuse of alcohol and active drugs within 12 months, except for nicotine; severe aphasia, visual and hearing impairment, etc. unable to complete the scale evaluation; MECT treatment contraindications; pregnant, lactating women or planning pregnancy; allergic to propofol and succinylcholine chloride.
  Interventions: Procedure: modified electroconvulsive therapy

INTERVENTIONS:
Procedure: modified electroconvulsive therapy — The patient underwent MECT therapy. The treatment instrument is Xingmaitong IV ECT multifunctional treatment instrument (USA, SOMATICS THYMATRON company), fasting for 6 hours before surgery, emptying urine. Routine preoperative preparations were made, followed by intravenous injection of atropine, propofol, and succinylcholine chloride injection, artificial respiration, placement of dental pads, and electroconvulsive therapy. The whole process is completed by an anesthesiologist and a therapist in cooperation with each other. The first 3 times are once a day, and the next 5 times are once every other day. A total of 8 courses of treatment.

SUMMARY:
To compare the correlation between the clinical efficacy of MECT treatment and baseline, 3 times, 8 times of treatment, 1 week after treatment, and 2 weeks after treatment in patients with depression and suicidal ideation. The prediction effect of -1β and IL-6 levels and level changes on the efficacy of MECT in the treatment of suicidal ideation in elderly patients with depression, and provide a theoretical basis for further research on the mechanism of MECT in the treatment of elderly depression with suicidal ideation.

DETAILED DESCRIPTION:
Late-life depression is a common mental disorder, old age 40-70% of the patients with suicide ideation, modified electroconvulsive therapy can quickly improve part in elderly patients with depression commit suicide idea, but curative effect exist individual differences, looking for MECT treatment of elderly patients with depression, early predictors of treatment plan formulation has important clinical significance.A total of 72 elderly patients with depression with suicidal thoughts were included in this project, who were treated with MECT for 8 times. Blood samples, demographic data and clinical symptom assessment data were collected before treatment, 3 times, 8 times, 1 week and 2 weeks after treatment, and the levels of IL-1β and IL-6 were measured at each time point. To analyze the relationship between the levels of IL-1β and IL-6 at baseline and at each time point and the changes of clinical symptoms and suicide concept, and to explore the predictive effect of the levels and changes of IL-1β and IL-6 on the efficacy of MECT in the treatment of suicide concept in elderly patients with depression. To provide a reference for further research on the mechanism of MECT in the treatment of senile depression with suicide.

ELIGIBILITY:
Inclusion Criteria:

Provide written informed consent; Age 60 to 85 years old, including 60 and 85 years old;

Meet the diagnostic criteria for single or recurrent major depressive disorder in DSM-5 (Diagnostic and Statistical Manual of Mental Disorders, 5th Edition);

Currently in the acute phase, with a total score of 17-item Hamilton Depression Rating Scale (HDRS-17) ≥ 24 at baseline;

History of suicide attempt in this depressive episode; Rating Scale (SIOSS)≥12 points;

Exclusion Criteria:

Patients with a history of epilepsy or coronary heart disease or other serious unstable physical diseases;

Patients with acute inflammatory infection or chronic inflammatory disease; Patients in the past 1 month Participated in another interventional clinical study;

Past or current diagnosis of the following psychiatric diseases by DSM-IV: organic mental disorder, Alzheimer's disease, secondary dementia due to other causes, mental illness Schizophrenia, schizoaffective disorder, bipolar disorder, delusional disorder, unspecified mental illness, and patients with a history of drug abuse, including alcohol and active drug abuse in the past 12 months, except for nicotine;

Severe aphasia , visual and hearing impairment, etc. who cannot complete the scale evaluation;

Those who have contraindications to MECT treatment;

Those who are pregnant, lactating women or planning to become pregnant; Those who are allergic to atropine, propofol, and succinylcholine chloride.

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All subjects were from elderly patients with depression who were hospitalized in Beijing Anding Hospital Affiliated to Capital Medical University.
Sampling Method: Non-Probability Sample
Enrollment: 72 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-10-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Change level of IL-6 compared with baseline at the end of MECT treatment. | baseline;through treatment 3 times, an average of 3 day;through treatment 8 times, an average of two weeks; three weeks;four weeks
  Serum IL-6 levels were measured at baseline, 3 times of treatment, 8 times of treatment, 1 week of treatment and 2 weeks of treatment. At the same time, SIOSS, BSI-CV, HDRS-17 and MADRS were used to comprehensively evaluate the clinical symptoms of elderly patients with depression.

SECONDARY OUTCOMES:
Change level of IL-1β compared with baseline at the end of MECT treatment. | baseline;through treatment 3 times, an average of 3 day;through treatment 8 times, an average of two weeks; three weeks;four weeks
  Serum IL-1β levels were measured at baseline, 3 times of treatment, 8 times of treatment, 1 week of treatment and 2 weeks of treatment. At the same time, SIOSS, BSI-CV, HDRS-17 and MADRS were used to comprehensively evaluate the clinical symptoms of elderly patients with depression.

CONTACTS AND LOCATIONS:
Overall Officials: Qing e Zhang, PhD, Study Chair — Beijing Anding Hospital Affiliated to Capital Medical University
Locations (1):
- Beijing Anding Hospital Affiliated to Capital Medical University, Beijing, Beijing Municipality, China

REFERENCES:
- [Result] Liu J, Yan F, Ma X, Guo HL, Tang YL, Rakofsky JJ, Wu XM, Li XQ, Zhu H, Guo XB, Yang Y, Li P, Cao XD, Li HY, Li ZB, Wang P, Xu QY. Prevalence of major depressive disorder and socio-demographic correlates: Results of a representative household epidemiological survey in Beijing, China. J Affect Disord. 2015 Jul 1;179:74-81. doi: 10.1016/j.jad.2015.03.009. Epub 2015 Mar 14. PMID 25845752
- [Result] Guerra M, Prina AM, Ferri CP, Acosta D, Gallardo S, Huang Y, Jacob KS, Jimenez-Velazquez IZ, Llibre Rodriguez JJ, Liu Z, Salas A, Sosa AL, Williams JD, Uwakwe R, Prince M. A comparative cross-cultural study of the prevalence of late life depression in low and middle income countries. J Affect Disord. 2016 Jan 15;190:362-368. doi: 10.1016/j.jad.2015.09.004. Epub 2015 Oct 23. PMID 26544620
- [Result] Carlier A, van Exel E, Dols A, Bouckaert F, Sienaert P, Ten Kate M, Wattjes MP, Vandenbulcke M, Stek ML, Rhebergen D. The course of apathy in late-life depression treated with electroconvulsive therapy; a prospective cohort study. Int J Geriatr Psychiatry. 2018 May 30. doi: 10.1002/gps.4917. Online ahead of print. PMID 29851173
- [Result] Obbels J, Verwijk E, Vansteelandt K, Dols A, Bouckaert F, Schouws S, Vandenbulcke M, Emsell L, Stek M, Sienaert P. Long-term neurocognitive functioning after electroconvulsive therapy in patients with late-life depression. Acta Psychiatr Scand. 2018 Sep;138(3):223-231. doi: 10.1111/acps.12942. Epub 2018 Jul 12. PMID 30003550